CLINICAL TRIAL: NCT05010733
Title: SPECT-CT Metabolic and Morphological Study of Two Types of Cemented Hip Stem Protheses in Primary Total Hip Arthroplasty Patients: A Randomized Controlled Clinical Trial (SPECT-PROTMA)
Brief Title: SPECT-CT Metabolic/Morphological Assessment of Cemented Hip Protheses
Acronym: SPECT-PROTMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daniel Rodriguez Perez (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Institut Català de la Salut (Other)
Responsible Party: Sponsor-Investigator, Daniel Rodriguez Perez, Principal Investigator, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUB- COT-2020-01
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Arthropathy of Hip
Keywords: Hip Arthroplasty; French Paradox; Thick-layer; SPECT; Metabolic changes; CT scan; Morphological changes

STUDY DESIGN:
Intervention Model Description: An anonymized list will be provided to the Biostatistics Department, who will randomly assign patients to a type of surgical intervention using a computer-generated randomization sequence. The randomization will be carried out previously to the surgery based on REDCap systems.
Masking Description: After assignment to interventions (Exeter V40 cemented femoral stem or Müller THA), participant and surgeon team will be aware of the type of cemented stem prosthesis allocated. Since after randomization this is an open-label study, emergency unblinding does not apply. Data analysts will be blinded.
  Personal patient data will be coded and dissociated, so that the patient to whom they correspond is not recognizable. Consecutive numbers will be assigned as they are enrolled in the study, and these numbers (or codes) will be used in the eCRF, rather than personal data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thick-Layer Technique (Experimental): Total hip arthroplasty using the Exeter V40 cemented femoral stem [Stryker Orthopaedics, Mahwah, New Jersey].
  Interventions: Device: Total hip arthroplasty using the Exeter V40 cemented femoral stem
- Thin-Layer Technique (French Paradox) (Active Comparator): Total hip arthroplasty using the Müller Straight Stem [Zimmer, Winterthur, Switzerland].
  Interventions: Device: Total hip arthroplasty using the Müller Straight Stem

INTERVENTIONS:
Device: Total hip arthroplasty using the Exeter V40 cemented femoral stem — Consists of applying a cement layer of at least 2 millimeters surrounding an undersized prosthetic stem, so that this layer of cement fits between the femoral medullary canal and the prosthetic's femoral stem.
  Other Names: Total hip arthroplasty using the Thick-Layer Technique
  Arms: Thick-Layer Technique
Device: Total hip arthroplasty using the Müller Straight Stem — Consists of applying a thin layer of cement, so that the prosthetic's femoral stem fills as much as possible the femoral medullary canal.
  Other Names: Total hip arthroplasty using the Thin-Layer Technique (French Paradox)
  Arms: Thin-Layer Technique (French Paradox)

SUMMARY:
Single center, pilot, randomized, controlled clinical trial to assess metabolic and morphological images between two types of cemented stem prostheses in patients undergoing total hip arthroplasty surgery during a 2-year follow up period.

DETAILED DESCRIPTION:
Single center, pilot, controlled clinical trial to assess metabolic and morphological images of patients undergoing total hip arthroplasty surgery randomized to the thick layer technique (Exeter hip stem model) or to the "French paradox" technique (Müller straight stem model).

Participants will be performed a plain radiography and a SPECT-CT at 3, 6, 12 and 24 months of the intervention. SPECT-CTs will be performed in addition to the usual medical care complementary imaging exams. The SPECT will require the administration of the 99mTechnetium-methylene diphosphonate (99mTc-MDP) radiopharmaceutical (useful to assess bone metabolism) and its combination with a CT scan (SPECT-CT) allows a combined metabolic and morphological study.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years-old
* both genders
* patients undergoing a primary total hip arthroplasty surgery with implantation of a cemented prosthesis (Exeter hip stem model or Müller straight stem model)
* patients with a diagnosis of hip osteoarthritis, operated by the Orthopedic Surgery and Traumatology Department at the Bellvitge University Hospital
* patients who signed the written informed consent.

Exclusion Criteria:

* patients allergic to 99mTc-MDP radiopharmaceutical
* patients with claustrophobia
* patients with a background of an active septic process
* patients with a postoperative septic complication
* patients periprosthetic fracture or misalignment of the prosthetic component
* patients who have a total hip prosthetic implanted due to a subcapital femoral fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of counts per image set in the SPECT study | 24 months after surgery
  Counts per image: unit of measure defined as the number of photons captured by the gamma camera, which represent the radiopharmaceutical uptake
Alignment angles in the plain radiography and in the CT scan study. | 24 months after surgery

SECONDARY OUTCOMES:
Axial displacement in the plain radiography and in the CT Scan study. | 24 months after surgery
Harris Radiographic Classification of Loosening Risk. | 24 months after surgery
Harris Hip Score | 24 months after surgery
Merle d'Aubigné Score | 24 months after surgery
WOMAC Index Score | 24 months after surgery
EuroQoL-5D-3L questionnaire score | 24 months after surgery
  Permission for this instruments' use has been granted by the EuroQoL Office.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Pérez, MD, Principal Investigator — Orthopedic Surgeon Specialized in Hip Arthroplasty
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holzwarth U, Cotogno G; Total hip arthroplasty: State of the art, prospects and challenges. EUR 25378 EN. Luxembourg (Luxembourg): Publications Office of the European Union; 2012. JRC72428
- [Background] Lopez franco, M. P. Yendo al hospital. Diagnóstico por la imagen. Sociedad Española de Proteccion Radiológica 2006.
- [Result] Brix G, Nekolla EA, Borowski M, Nosske D. Radiation risk and protection of patients in clinical SPECT/CT. Eur J Nucl Med Mol Imaging. 2014 May;41 Suppl 1:S125-36. doi: 10.1007/s00259-013-2543-3. Epub 2013 Sep 20. PMID 24052089
- [Result] El Masri F, Kerboull L, Kerboull M, Courpied JP, Hamadouche M. Is the so-called 'French paradox' a reality?: long-term survival and migration of the Charnley-Kerboull stem cemented line-to-line. J Bone Joint Surg Br. 2010 Mar;92(3):342-8. doi: 10.1302/0301-620X.92B3.23151. PMID 20190303
- [Result] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Result] Harris WH, McCarthy JC Jr, O'Neill DA. Femoral component loosening using contemporary techniques of femoral cement fixation. J Bone Joint Surg Am. 1982 Sep;64(7):1063-7. PMID 7118973
- [Result] Harris WH. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. J Bone Joint Surg Am. 1969 Jun;51(4):737-55. No abstract available. PMID 5783851
- [Result] Merle D'Aubigne R. [Numerical classification of the function of the hip. 1970]. Rev Chir Orthop Reparatrice Appar Mot. 1990;76(6):371-4. No abstract available. French. PMID 2149773
- [Result] Mushtaq N, To K, Gooding C, Khan W. Radiological Imaging Evaluation of the Failing Total Hip Replacement. Front Surg. 2019 Jun 18;6:35. doi: 10.3389/fsurg.2019.00035. eCollection 2019. PMID 31275942
- [Result] Ovre S, Sandvik L, Madsen JE, Roise O. Comparison of distribution, agreement and correlation between the original and modified Merle d'Aubigne-Postel Score and the Harris Hip Score after acetabular fracture treatment: moderate agreement, high ceiling effect and excellent correlation in 450 patients. Acta Orthop. 2005 Dec;76(6):796-802. doi: 10.1080/17453670510045390. PMID 16470432
- [Result] Roos EM, Klassbo M, Lohmander LS. WOMAC osteoarthritis index. Reliability, validity, and responsiveness in patients with arthroscopically assessed osteoarthritis. Western Ontario and MacMaster Universities. Scand J Rheumatol. 1999;28(4):210-5. doi: 10.1080/03009749950155562. PMID 10503556
- [Result] Son HJ, Jeong YJ, Yoon HJ, Wang L, Kim HJ, Park JH, Kang DY. Visual Pattern and Serial Quantitation of 18F-Sodium Fluoride PET/CT in Asymptomatic Patients After Hip and Knee Arthroplasty. Nucl Med Mol Imaging. 2016 Dec;50(4):308-321. doi: 10.1007/s13139-016-0430-0. Epub 2016 Jul 13. PMID 27994686
- [Result] Tam HH, Bhaludin B, Rahman F, Weller A, Ejindu V, Parthipun A. SPECT-CT in total hip arthroplasty. Clin Radiol. 2014 Jan;69(1):82-95. doi: 10.1016/j.crad.2013.08.003. Epub 2013 Sep 15. PMID 24047953
- [Result] Van den Wyngaert T, Strobel K, Kampen WU, Kuwert T, van der Bruggen W, Mohan HK, Gnanasegaran G, Delgado-Bolton R, Weber WA, Beheshti M, Langsteger W, Giammarile F, Mottaghy FM, Paycha F; EANM Bone & Joint Committee and the Oncology Committee. The EANM practice guidelines for bone scintigraphy. Eur J Nucl Med Mol Imaging. 2016 Aug;43(9):1723-38. doi: 10.1007/s00259-016-3415-4. Epub 2016 Jun 4. PMID 27262701
- [Result] Venesmaa P, Vanninen E, Miettinen H, Kroger H. Periprosthetic bone turnover after primary total hip arthroplasty measured by single-photon emission computed tomography. Scand J Surg. 2012;101(4):241-8. doi: 10.1177/145749691210100404. PMID 23238498
- [Result] Yamane T, Kuji I, Seto A, Matsunari I. Quantification of osteoblastic activity in epiphyseal growth plates by quantitative bone SPECT/CT. Skeletal Radiol. 2018 Jun;47(6):805-810. doi: 10.1007/s00256-017-2861-9. Epub 2018 Jan 11. PMID 29327129
- [Result] Yang Z, Reed T, Longino BH. Bone Scintigraphy SPECT/CT Evaluation of Mandibular Condylar Hyperplasia. J Nucl Med Technol. 2016 Mar;44(1):49-51. doi: 10.2967/jnmt.115.158691. Epub 2015 Jun 25. PMID 26111714
- [Derived] Rodriguez D, Carnaval T, Del Carmen M, Palomar-Munoz A, Cortes-Romera M, Agullo JL, Videla S. SPECT-CT metabolic and morphological study of 2 types of cemented hip stem prostheses in primary total hip arthroplasty patients: A protocol for a randomized controlled clinical trial (SPECT-PROTMA). Medicine (Baltimore). 2021 Dec 30;100(52):e28299. doi: 10.1097/MD.0000000000028299. PMID 34967362
- See also: Lopez franco, M. P. Yendo al hospital. Diagnóstico por la imagen. Sociedad Española de Proteccion Radiológica 2006. — https://www.sepr.es/profesionales/descargables/download/82-area-medica/4070-yendo-al-hospital-i-diagnostico-por-imagen-radiodiagnostico-y-medicina-nuclear
- See also: Holzwarth U, Cotogno G; Total hip arthroplasty: State of the art, prospects and challenges. EUR 25378 EN. Luxembourg (Luxembourg): Publications Office of the European Union; 2012. JRC72428 — https://publications.jrc.ec.europa.eu/repository/handle/JRC72428